CLINICAL TRIAL: NCT06263062
Title: Impact of the Awareness-Based Initiation Program on Cancer Fear and Awareness Level in Women Undergoing Colposcopy: Randomized Controlled Study
Brief Title: Management With Fear of Cancer in Women Undergoing Colposcopy: Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Fatma Ozlem Uner, Research Assistant, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: women undergoing colposcopy
Record Dates: First submitted 2024-02-07; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Cancer Fear; Cervical Cancer
Keywords: fear of cancer; MBSR; nursing; awareness; cervical cancer
MeSH Terms: conditions — Pathophobia; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): routine care after a colopscopy procedure "Mindfulness-Based Coping Programme" in addition to routine care Prepared in accordance with the MBSR programme. Applied online with Zoom programme Teams in groups of 6 people 6 sessions in 2 weeks
  Interventions: Behavioral: Awareness-Based Coping with Fear of Cancer Programme
- Control group (No Intervention): routine care after a colopscopy procedure Routine care will be provided by the nurse training handbook created by the researcher

INTERVENTIONS:
Behavioral: Awareness-Based Coping with Fear of Cancer Programme — The content of the Training Program was created by researchers based on MBSR, in line with high-level research results and international guides.Then, the necessary arrangements were made bytaking the opinions of 10 experts ( faculty members of the department of obstetrics and gynaecology nursing, psychiatry specialist, faculty members of the gynaecology oncology department, oncology clinic psychologist, obstetrics and gynaecology clinic charge nurse). Content concluded in accordance with the comments received.
  Arms: Experimental group

SUMMARY:
Cervical cancer is the fourth most common cancer in women worldwide. Due to advances in early diagnosis and treatment, the number of survivors of cancer has increased over the past 50 years. Therefore, the current standard of care for the detection of cervical neoplasm, a Papanicolaou smear and then a colposcopic biopsy, requires a high degree of diagnostic accuracy. In particular, the fear of developing cancer after cancer screening tests is becoming an increasingly significant problem, with an impact on psychosocial health in individuals. For people who are afraid of cancer, meditation and awareness training can make it easier for emotions to self-regulate in times of distress and pain. This study aim to conducted to determine the impact of the Awareness-Based Initiation Program on cancer fear and level of awareness in women undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Colposcopy procedure due to HSIL, LSIL, ASC-H or HPV on cervical cytology
* Volunteering to participate in the 6-session Mindfulness-Based Coping Programme Knowing what a colposcopy procedure means,

Exclusion Criteria:

* interference with verbal communication,
* being diagnosed with major depressive disorder or psychiatric disorder,
* having participated in MBSR training or meditating before
* Lack of skills to use smart phones and computers
* learning biopsy results during the programme

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Enrollment: 60 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
The Cancer Worry Scale | This scale will be administered twice: pre-intervention and immediately after the intervention
  The Cancer Worry Scale was developed by Custers et al. (2014) and consists of 8 items. In the Likert scale, the responses are numbered from 0 to 4. In the scale, 0 is expressed as "almost never", while 4 is expressed as "almost always". In the scoring of the scale, the lowest score is 0 and the highest score is 32. Cronbach's alpha value was determined as 0.87.

SECONDARY OUTCOMES:
Philadelphia Mindfulness Scale | This scale will be administered twice: pre-intervention and immediately after the intervention
  Philadelphia Mindfulness Scale The scale developed by Cardaciotto et al. in 2008 is a five-point Likert-type scale consisting of 20 items. The scale measures awareness skills in two different dimensions: (i) discrimination (awareness), (ii) acceptance (acceptance). In the original validity and reliability study of the scale, Cronbach's alpha value was determined as 0.85. The two sub-dimensions of the scale were determined as discrimination (α=.81) and acceptance subscale (α=.86).

CONTACTS AND LOCATIONS:
Overall Officials: fatma ozlem uner, MSc, Principal Investigator — Alanya Alaaddin Keykubat University
Locations (1):
- Alanya Alaaddin Keykubat University, Alanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No